CLINICAL TRIAL: NCT06709027
Title: The Construction and Application of a Mobile Health Management Program for Elderly Depression Based on the Patterns of Cognitive Function Changes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Zhu Ziping, Fujian Medical University, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-87; 2018-87 (Other: FujianMU)
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Patients With Depression in the Elderly

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment design where participants are randomly assigned to either the experimental group receiving Mobile Health Management Intervention or the control group receiving a standard treatment. The study is single-blind, meaning participants are unaware of which group they belong to, thus minimizing potential bias. Data will be collected at regular intervals to evaluate the efficacy and safety of the intervention.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Mobile Health Management Intervention) (Experimental): Participants in this group will receive a mobile health management intervention over a period of 12 weeks. This intervention includes the use of a mobile application designed for health management, psychological support, and monitoring，et al, with the aim of improving the mental health status of elderly patients with depression.
  Interventions: Device: Intervention Group (Mobile Health Management Intervention)
- Control Group (Standard Care) (No Intervention): Participants in this group will receive standard care during the same 12-week period. This includes routine medical services and psychological support, but does not involve any specific mobile health intervention.

INTERVENTIONS:
Device: Intervention Group (Mobile Health Management Intervention) — Participants in this group will receive a mobile health management intervention over a period of 12 weeks. This intervention includes the use of a mobile application designed for health management, psychological support, and monitoring,et al， with the aim of improving the mental health status of elderly patients with depression.
  Arms: Intervention Group (Mobile Health Management Intervention)

SUMMARY:
Based on the changing law of cognitive function, combined with the behavior change wheel theory and the health behavior process orientation model, we constructed a mobile health management program for geriatric depression. The aim is to explore the effect of this intervention program on the health behavior of elderly patients with depression; and to verify the effect of the intervention program on improving the primary outcome and other secondary outcomes of elderly patients with depression, with a view to providing a scientific basis for the management of depression in the elderly and promoting the optimization of personalized intervention strategies.

DETAILED DESCRIPTION:
Based on the changing law of cognitive function, combined with the behavior change wheel theory and the health behavior process orientation model, we constructed a mobile health management program for geriatric depression. The aim is to explore the effect of this intervention program on the health behavior of elderly patients with depression; and to verify the effect of the intervention program on improving the primary outcome and other secondary outcomes of elderly patients with depression, with a view to providing a scientific basis for the management of depression in the elderly and promoting the optimization of personalized intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* ① Meet the clinical diagnosis of geriatric depression and DSM-5 diagnostic criteria; ② Age ≥ 60 years old, clear consciousness; ③ Be able to communicate in Mandarin, with a certain degree of comprehension and expression; ④ Possess a smart phone and have the ability to operate it in a basic way; ⑤ Voluntarily participate in this study and sign an informed consent form

Exclusion Criteria:

* ①previous or current cognitive impairment and other severe mental illnesses that prevent cooperation with the study;②comorbidities such as severe cardiac, hepatic, or renal impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
cognitive function | From baseline (T0) to 6 weeks post-intervention (T1) and 12 weeks post-intervention (T2)
  Using Montreal Cognitive Assessment（ MoCA） to assess patients' cognitive function

SECONDARY OUTCOMES:
depressive symptoms | From baseline (T0) to 6 weeks post-intervention (T1) and 12 weeks post-intervention (T2)
  sing the Geriatric Depression Scale (GDS-15) to assess patients' depressive symptoms.
Behavioral Inhibition /Behavioral Activation | From baseline (T0) to 6 weeks post-intervention (T1) and 12 weeks post-intervention (T2)
  Using the Behavioral Inhibition System/Behavioral Activation System Scale (BIS/BAS) to assess patients' behavior.
patients' quality of life | From baseline (T0) to 6 weeks post-intervention (T1) and 12 weeks post-intervention (T2)
  Using the WHO QOL-BREF to assess patients' quality of life.
sleep quality | From baseline (T0) to 6 weeks post-intervention (T1) and 12 weeks post-intervention (T2)
  Using the Pittsburgh Sleep Quality Index (PSQI) to assess patients' sleep quality.
psychological needs | From baseline (T0) to 6 weeks post-intervention (T1) and 12 weeks post-intervention (T2)
  Using the Basic Psychological Needs Scale (BPNS) to assess patients' psychological needs.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medial University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
2025.7.1
Supporting Information: Study Protocol